CLINICAL TRIAL: NCT00404664
Title: A Novel Approach To Improve Influenza Vaccination Rates Among Health Care Professionals: A Prospective Randomized Controlled Trial
Brief Title: Improving Influenza Vaccination Rates Among Health Care Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: IRB 7370
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Influenza
Keywords: influenza vaccine; influenza immunization; reminder letters; raffle prize
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Behavioral: influenza vaccine, reminders letters, raffle prize

SUMMARY:
The purpose of this study was to see if reminder letters and a large raffle prize would encourage health care workers to receive influenza vaccinations.

DETAILED DESCRIPTION:
Eight hundred employees of an urban tertiary care hospital, 200 each from the following four categories: professional staff, resident physicians, registered nurses, and licensed practical nurses comprised the study group. Subjects were randomly assigned to receive: 1) no intervention, 2) a reminder letter for flu vaccine, 3) a raffle ticket to win a free Caribbean vacation with flu vaccine administration, or 4) both the reminder letter and raffle ticket. We compared the proportion of employees receiving vaccination and participating in the raffle across groups.

ELIGIBILITY:
Inclusion Criteria:

* Hospital employees, staff physicians, residents, rn's, lpn's

Exclusion Criteria:

* non patient care hospital employees

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800
Dates: Start 2004-09; Study Completion 2005-04

PRIMARY OUTCOMES:
Proportion of employees receiving vaccination and participating in the raffle across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Macknin, M.D., Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States